CLINICAL TRIAL: NCT03996980
Title: Effect Mechanism of Custom-made Foot Orthoses on Foot Pronation Subjects and Chronic Low Back Pain: a Randomized Controlled Trial
Brief Title: Effect Mechanism of Custom-made Foot Orthoses in Patients With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, MANUEL PABON CARRASCO, Principal Investigator, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRESEUE-Foot
Record Dates: First submitted 2019-06-09; First posted 2019-06-25 (Actual); Results first posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2024-05

CONDITIONS: Chronic Low Back Pain; Foot Pronation
Keywords: Low back pain; custom-made foot orthoses; Foot; pronation; posture
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Custom-made foot orthoses (Experimental): treatment intervention custom-made polypropylene foot orthoses for a period of 4 weeks
  Interventions: Device: Custom-made foot orthoses Versus a flat insole
- Placebo (Placebo Comparator): a flat insole for a period of 4 weeks
  Interventions: Device: Custom-made foot orthoses Versus a flat insole

INTERVENTIONS:
Device: Custom-made foot orthoses Versus a flat insole — Compare the use of plantar orthoses (experimental group) with the use of a flat insoles (control group)

SUMMARY:
Excessive foot pronation has been recognized as being linked to chronic low back pain (CLBP). The use of compensating custom-made foot orthoses has not been entirely explored as an effective therapy for CLBP Objective: to investigate the effects of wearing custom made foot orthoses compared to placebo orthoses in patients with pronated feet and chronic low back pain (CLBP).

DETAILED DESCRIPTION:
Excessive foot pronation has been recognized as being linked to CLBP. Foot hyperpronation may cause malalignment of the lower extremity.There is a wide variety of treatments for CLBP, and it is suggested that excessive pronation of the foot has been linked to CLBP.The use of compensating custom-made foot orthoses has not been entirely explored as an effective therapy for CLBP.

Customized foot orthoses alter the position of the foot during weight-bearing. The goal is to eliminate compensation of the foot due to structural deformity or misalignment and redistribute abnormal plantar pressures.Custom-made foot orthoses may contribute to improving chronic low back pain. This question represents an important benefit for patients and for the public health system by reducing expensive treatments, such as surgery or long periods of rehabilitation

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 18 and 65 years old
* Presence of CLBP
* Foot Posture Index pronated in one or both feet (henceforth, FPI) ≥ +6

Exclusion Criteria:

* Serious illness
* Current participation in another research study
* Pregnancy
* Previous back or foot surgery
* Current treatment of foot pathology or back, and leg length discrepancy > 5 mm

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2013-01-15 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-07-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - university. Departament of Podiatry, Seville
  - Manuel Pabón Carrasco, Seville

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: . The random allocation to each group was done by a collaborating researcher who established the sequence based on a random numbers table and then the treatment was administered (experimental/control).
Pre-assignment Details: Participants are excluded if they have a pregnancy during the study. Pregnancy modifies the curvature of the back.
  All those processes that alter the physiology of the musculoskeletal system will also be excluded.
Period: Overall Study
Arm/Group | Custom-made Foot Orthoses | Placebo
Started | 55 | 55
Completed | 53 | 48
Not Completed | 2 | 7

BASELINE CHARACTERISTICS:
Population: 101 patients with nonspecific CLBP and a pronated foot posture index (FPI) was studied. Randomized in two groups, an experimental one n= 53, used custom-made foot orthotics and the control group n=48 treated with non-biomechanical effect orthoses
Groups:
- Total: Total of all reporting groups
Arm/Group | Custom-made Foot Orthoses | Placebo | Total
Number analyzed (Participants) | 53 | 48 | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 53 | 48 | 101
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 28 | 56
  Male | 25 | 20 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 53 | 48 | 101
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Oswestry's Disability Index Questionnaire [Mean (Standard Deviation); unit: units on a scale Minimum 0% Maximum 100] — 0% to 20%: minimal disability 21%-40%: moderate disability 41%-60%: severe disability. 61%-80%: crippled 81%-100%: These patients are either bed-bound or exaggerating their symptoms.
  units on a scale Minimum 0% Maximum 100 | 20.45 (1.7) | 19.02 (1.37) | 20 (1.6)
visual analogue scale (VAS) [Median (Standard Deviation); unit: units on a scale Minimum 0 Maximum 10] — no pain (0-2), mild pain(2-4), moderate pain (4-7), and severe pain (7-10)
  units on a scale Minimum 0 Maximum 10 | 6.36 (0.23) | 6.26 (0.25) | 6.30 (0.24)

OUTCOME MEASURES:

1. Primary Outcome: Oswestry Disability Index Questionnaire(ODI) for Lower Back Pain
Description: This questionnaire has been designed to give us information as to how your back or leg pain is affecting your ability to manage in everyday life.The test is considered the 'gold standard' of low back functional outcome tools 0% to 20%: minimal disability: The patient can cope with most living activities.
  21%-40%: moderate disability: The patient experiences more pain and difficulty with sitting, lifting and standing. Travel and social life are more difficult and they may be disabled from work. Personal care, sexual activity and sleeping are not grossly affected and the patient can usually be managed by conservative means. 41%-60%: severe disability: Pain remains the main problem in this group but activities of daily living are affected. These patients require a detailed investigation. 61%-80%: crippled: Back pain impinges on all aspects of the patient's life. Positive intervention is required. 81%-100%: These patients are either bed-bound or exaggerating their symptoms.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Score on 0-100% scale
Arm/Group | Custom-made Foot Orthoses | Placebo
Number analyzed (Participants) | 53 | 52
Score on 0-100% scale | 20.45 (12.51) | 19.02 (9.5)

2. Primary Outcome: VAS for Chronic Low Back Pain
Description: 10 visual analogue scale (VAS).The findings suggested that 10 VAS ratings of no pain (0-2), mild pain(2-4), moderate pain (4-7), and severe pain (7-10)
Time Frame: Baseline
Population: The groups are expected to be similar in gender, sex, age, pain at first (VAS and ODI) and at the time of the initial examination.This would allow a comparison avoiding risk of bias.
Measure: Mean (Standard Deviation); unit: Score on 0-10 scale
Arm/Group | Custom-made Foot Orthoses | Placebo
Number analyzed (Participants) | 53 | 48
Score on 0-10 scale | 6.36 (0.23) | 6.56 (0.24)

3. Primary Outcome: Foot Posture Index
Description: Foot posture was assessed by a podiatrist during the biomechanical assessment based on the six-item foot posture index (FPI≥+6). The FPI consists of six validated items that are measured in a relaxed standing position of the subject. Each item is assessed on a -2 to +2 scale, where -2 indicates a supinated position, 0 indicates a neutral position and +2 indicates a pronated position, depending on the specific item. The sum of the scores of the six items provides a total score ranging from -12 to +12.
Time Frame: At the moment of inclusion in the study
Measure: Mean (Standard Deviation); unit: Score on -12 to +12 scale
Arm/Group | Custom-made Foot Orthoses | Placebo
Number analyzed (Participants) | 53 | 48
Score on -12 to +12 scale | 5.98 (1.62) | 6.42 (1.33)

4. Secondary Outcome: Oswestry Disability Index Questionnaire (ODI)
Description: Oswestry Disability Index Questionnaire (ODI) for chronic low back pain
Time Frame: at the end of the study, approximately 4 weeks
Measure: Mean (Standard Deviation); unit: Score on 0-100% scale
Arm/Group | Custom-made Foot Orthoses | Placebo
Number analyzed (Participants) | 53 | 48
Score on 0-100% scale | 7.21 (6.20) | 21.17 (8.1)

5. Secondary Outcome: VAS
Description: VAS scale for CLBP
  Using a ruler, the score is determined by mea-suring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-10. A higher score indicates greater pain intensity.
Time Frame: At 4 weeks after baseline
Measure: Mean (Standard Deviation); unit: points on a 0-10 Visual Analogue Scale
Arm/Group | Custom-made Foot Orthoses | Placebo
Number analyzed (Participants) | 53 | 48
points on a 0-10 Visual Analogue Scale | 3.02 (1.80) | 6.54 (1.51)

ADVERSE EVENTS:
Time Frame: Adversor effects are valued for one months.
Description: The use of plantar supports does not result in participant mortality or serious adverse effects.
  Non-serious adverse effects are monitored.
Arm/Group | Custom-made Foot Orthoses | Placebo
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/52
Other Adverse Events (participants affected / at risk) | 0/53 | 0/52

LIMITATIONS AND CAVEATS:
The sample size should be expanded.

Treatment follow-up is difficult to assess (the patient goes home with treatment)

Future studies are necessary

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-04): https://cdn.clinicaltrials.gov/large-docs/80/NCT03996980/Prot_SAP_000.pdf